CLINICAL TRIAL: NCT06961422
Title: Impacts of Occupational Fatigue on the Mental Health of Shift Workers in Textile Industry of Karachi: A Cross-Sectional Study
Brief Title: Association Between Occupational Fatigue and Mental Health Among Textile Shift Workers in Pakistan
Status: Completed | Type: Observational
Sponsor: Rawalpindi Medical College (Other)
Responsible Party: Principal Investigator, Nazeer Ahmed, Final year medical student, Rawalpindi Medical College
Other Study IDs: approval number: PH-46-46-21
Record Dates: First submitted 2025-04-29; First posted 2025-05-08 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Occupational Diseases; Mental Disorders; Fatigue
Keywords: Occupational Fatigue; Shift Work; Mental Health; Textile Industry; Workplace Stress
MeSH Terms: conditions — Occupational Diseases; Mental Disorders; Fatigue; Psychological Well-Being; Occupational Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Brief Summary

The goal of this observational study is to evaluate how occupational fatigue affects mental health outcomes in adult shift workers employed in the textile industry. The main questions it aims to answer are:

What is the prevalence of mental health complaints among textile industry shift workers? How does occupational fatigue influence these mental health outcomes? Researchers will compare different levels of fatigue (based on MFI-20 scores) and their association with mental health status (based on GHQ-28 scores) to see if higher occupational fatigue is linked with poorer mental health.

Participants will:

Complete the Multidimensional Fatigue Inventory (MFI-20) to assess physical and mental fatigue.

Complete the General Health Questionnaire (GHQ-28) to screen for psychological distress.

Provide demographic and work-related information through a structured survey.

DETAILED DESCRIPTION:
Detailed Description

This study aims to assess the impact of occupational fatigue on the mental health of shift workers in the textile industry of Karachi. Given the growing concern about mental health issues in industries requiring extended hours and irregular shifts, this research seeks to identify how fatigue related to shift work affects the mental well-being of textile workers.

Study Design and Methodology

A cross-sectional study design will be employed to collect data from a sample of 356 shift workers in the textile sector. The sample will be selected using stratified random sampling to ensure a representative distribution across different demographic categories such as age, gender, and job type. Participants will be chosen from textile factories based in Karachi to provide a broader understanding of mental health issues in this sector.

Inclusion and Exclusion Criteria

The study will include workers who have been employed in the textile industry for at least six months. Workers with pre-existing mental health disorders, as identified by medical records, will be excluded to ensure the study focuses on occupational fatigue rather than underlying health conditions.

Data Collection Tools

Two standardized instruments will be used for data collection:

General Health Questionnaire (GHQ-28): This tool will assess the mental health status of participants, specifically focusing on symptoms such as anxiety, depression, and social dysfunction.

Multidimensional Fatigue Inventory (MFI-20): This will measure the severity of fatigue in the workers, evaluating both physical and mental fatigue, which may contribute to the workers' overall well-being.

Data will be gathered through face-to-face interviews and self-administered surveys. Informed consent will be obtained from each participant, ensuring that they understand the study's purpose and their right to confidentiality.

Statistical Analysis

The data will be analyzed using descriptive and inferential statistics. Descriptive statistics will summarize the demographic characteristics of the sample and the responses to the GHQ-28 and MFI-20. For inferential analysis, multiple regression analysis will be performed to explore the relationship between occupational fatigue and mental health, adjusting for potential confounders such as age, gender, and job type.

Ethical Considerations

The study has received ethical approval from the RSRS Ethical Review Board. All participants will provide written informed consent, and confidentiality will be maintained throughout the research process. The study will comply with ethical standards for research involving human subjects.

Expected Outcomes

The study is expected to find a significant correlation between occupational fatigue and poor mental health among shift workers. The findings could highlight the importance of fatigue management in improving the mental health of workers, suggesting the need for workplace interventions such as rest periods, psychological support programs, and changes in shift scheduling.

Limitations

This study is limited by its cross-sectional nature, which will only allow for the identification of associations rather than causal relationships. Additionally, the results may not be generalizable to workers in other industries or regions outside of Karachi.

ELIGIBILITY:
Inclusion Criteria:

* Workers employed in the textile industry for at least 6 months
* Involved in regular shift work (day/night rotation)
* Aged between 18 to 65 years
* Able to provide informed consent
* Willing to complete self-administered questionnaires

Exclusion Criteria:

* Diagnosed psychiatric disorders before employment
* Current use of psychotropic medications
* Diagnosed sleep disorders unrelated to occupational fatigue
* Severe physical illness or disability that may affect fatigue or mental health assessment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population includes male and female shift workers employed in textile industries, representing various departments (production, packaging, quality control, etc.), selected through stratified random sampling to ensure representation across shifts and job roles.
Sampling Method: Probability Sample
Enrollment: 356 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Assessment of Mental Health Status Using GHQ-28 | April 2023 to June 2024
  This outcome measures the mental health status of shift workers using the General Health Questionnaire-28 (GHQ-28). The tool evaluates four domains: somatic symptoms, anxiety and insomnia, social dysfunction, and severe depression. Scores help identify probable mental health issues among workers.

SECONDARY OUTCOMES:
Assessment of Occupational Fatigue Using Multidimensional Fatigue Inventory (MFI-20) | April 2023 to June 2024
  This outcome measures occupational fatigue among shift workers using the Multidimensional Fatigue Inventory (MFI-20). The tool assesses five domains: general fatigue, physical fatigue, mental fatigue, reduced activity, and reduced motivation. Higher scores indicate greater fatigue levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Textile Industry Workers' Health Research Center, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data (IPD) for this study, including demographic details and responses from the GHQ-28 and MFI-20 assessments, will be shared upon request. The data will be anonymized and de-identified to protect participants' confidentiality. The sharing will be done with researchers who wish to further analyze the impact of occupational fatigue and mental health in shift workers in textile industries.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The IPD and supporting information will be available for sharing starting from July 1025 and will remain available for 5 years (until January 2030).
Access Criteria: Researchers who submit a formal request and agree to a data-sharing agreement will be granted access to the IPD. They will be able to access de-identified individual-level data and the associated analytic code. The data will be shared through a secure online portal.

REFERENCES:
- Available data/document: Individual Participant Data Set: 0009-0009-61 — https://orcid.org/0009-0009-6142-6201